CLINICAL TRIAL: NCT02996656
Title: Antimicrobial Prophylaxis for Skin Colonization With Propionibacterium Acnes in Primary Open Shoulder Surgery: A Double Blinded Randomized Controlled Trial
Brief Title: Antimicrobial Prophylaxis for Skin Colonization With Propionibacterium Acnes in Primary Open Shoulder Surgery
Acronym: PAPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Stryker Trauma and Extremities (Industry); Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Dominique Rouleau, Orthopaedic surgeon, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PAPA
Record Dates: First submitted 2016-11-25; First posted 2016-12-19 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Propionibacterium Infection
MeSH Terms: interventions — Cefazolin; Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefazolin (Active Comparator): During an open shoulder surgery, the Cefazolin will be administered to some patient. The Cefazolin is a first generation cephalosporin. It is a beta lactam which targets gram positive cocci and some gram negative bacilli. The INESS Antibiotic Prophylaxis in Orthopedic Guide recommends the use of Cefazolin at induction for all orthopaedic procedure with implantation of internal fixation device. The dosage is 2g intravenous if the patient weights less than 120kg or 3g if the patient weights more than 120kg. The dose should be repeated if the procedure lasts for more than three hours or if the blood loss is greater than 1500mL.
  Interventions: Drug: Cefazolin
- Ceftriaxone (Experimental): During an open shoulder surgery, the Ceftriaxone will be administered to some patient. The Ceftriaxone is a third generation cephalosporin. It targets gram positive cocci such as staphylococcus and streptococcus, gram negative bacilli and some anaerobes, including P. acnes. The prophylactic dose is of 2g IV given a minimum of 30 minutes prior to skin incision. It is effective 12h so no other dose is needed during surgery.
  Interventions: Drug: Ceftriaxone

INTERVENTIONS:
Drug: Cefazolin — Antibiotic that will be give before a Trauma or elective open shoulder surgery
  Arms: Cefazolin
Drug: Ceftriaxone — Antibiotic that will be give before a Trauma or elective open shoulder surgery
  Arms: Ceftriaxone

SUMMARY:
INESS Antibiotic Prophylaxis in Orthopedic Guide recommends the use of Cefazolin at induction for all orthopaedic procedure with implantation of internal fixation device. With the increasing rate of identified P. acnes shoulder surgery infection despite the use of recommended skin preparation and preoperative prophylactic antibiotics, a question arises; Is Cefazolin the most effective prophylactic antibiotic for shoulder surgery? The objective of this study is to determine if Ceftriaxone is superior to Cefazolin as a prophylactic antibiotic for skin colonization with P. acnes in primary shoulder surgery

DETAILED DESCRIPTION:
This is a double blinded randomized clinical trial comparing two different prophylactic antibiotics used for primary open shoulder surgery. The participants are volunteer patients scheduled for a primary open elective or trauma shoulder surgery. Patients with positive MRSA screening test will be excluded from the randomised study as they will receive vancomycin for prophylaxis. If they accept to participate, they will be included in the observational MRSA+ arm. The investigators will take from the participants the same data as the randomised patients and the investigators will take biopsies.

4 equals group will be form: Female-elective: 22 envelops, 11 cefazolin, 11 ceftriaxone in a randomly order Female-trauma: 22 envelops, 11 cefazolin, 11 ceftriaxone in a randomly order Male-elective: 22 envelops, 11 cefazolin, 11 ceftriaxone in a randomly order Male-trauma: 22 envelops, 11 cefazolin, 11 ceftriaxone in a randomly order The surgeons, anesthesiologist, patients and laboratory technician, microbiologist will be blinded to the antibiotics received by the patient.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Male or female
* Presenting normal skin on the shoulder aria

Exclusion Criteria:

* Used antibiotics or treated their skin with antibiotic gel, alcohol gel or cream or acne treatment in the last three months
* Active infection at the surgical site or anywhere
* Affected shoulder previously received radiotherapy
* Allergic to one of the antimicrobial prophylaxis used
* Open fracture
* Life threatening or a limb threatening pathology
* Liver or kidney failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2016-12; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Skin Biopsy | At the initial surgery
  Number of bacteria identified in five skin biopsies taken at the surgical site

SECONDARY OUTCOMES:
MRSA observance | 1 year following the surgery
  Observe the patients from de MRSA group which will be receiving Vancomycin as prophylactic antibiotics.
Infection | 1 year following the surgery
  Assessing the appearance of C Difficile infection at 1 year post-op
Infection #2 | 1 year following the surgery
  Assessing the appearance of resistant pathogens colonization (MRSA, VRE, Multiresistant Gram negative Bacillus) 1 year post-op
Infection #3 | 1 year following the surgery
  Follow all the participants for one year to observe superficial tissue infection (as defined by the infection prevention team of Montreal Sacre-Coeur Hospital
Infection #4 | 1 year following the surgery
  Follow all the participants for one year to observe deep tissue infection (as defined by the infection prevention team of Montreal Sacre-Coeur Hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Rouleau, MD, Principal Investigator — Université de Montréal
Locations (1):
- Hôpital du Sacré-Cœur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided